CLINICAL TRIAL: NCT04436809
Title: Sentinel Node Biopsy Alone or With Axillary Dissection in cT2 cN0/1 Breast Cancer Patients After Primary Chemotherapy: a Prospective Interventional Study
Brief Title: Sentinel Node Biopsy Alone or With Axillary Dissection After Primary Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Gabriele Martelli, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT180/13
Record Dates: First submitted 2020-06-14; First posted 2020-06-18 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Breast Neoplasm Female
Keywords: Breast cancer; Sentinel node biopsy; Neoadjuvant chemotherapy; Axillary dissection
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNB only (Other): cT2 patients scheduled for primary chemotherapy (with or without a clinically involved axilla - cN0/1) who have disease-free sentinel nodes (pN0) after primary chemotherapy, are directed to "SNB only": i.e. no further treatment to the axilla.
  Interventions: Procedure: Sentinel Node Biopsy
- SNB + AD (Other): cT2 patients scheduled for primary chemotherapy (with or without a clinically involved axilla - cN0/1) who have metastatic sentinel nodes (pN1) on sentinel node biopsy (SNB) will undergo axillary dissection (AD) i.e. surgical removal of most axillary lymph nodes.
  Interventions: Procedure: Sentinel Node Biopsy; Procedure: Axillary Dissection

INTERVENTIONS:
Procedure: Sentinel Node Biopsy — Colloidal radiotracer (99Tc) is injected into the breast near the cancer. The radiotracer moves in the lymph ducts to accumulate in the first lymph nodes (almost always in the axilla) to receive lymph from the breast area containing the cancer. Lymphoscintigraphy is used to check for the presence of radioactivity in the axilla. Some hours later, during breast surgery, a radioactivity-detecting probe is used to identify "hot" lymph nodes (sentinel nodes) and aid their surgical removal from the axilla. These nodes are examined histologically (intraoperatively) for the presence of cancer. If they are disease-free the axilla will be left intact (no further axillary treatment given); if they contain cancer most lymph nodes in the axilla will be removed surgically (axillary dissection).
  Other Names: Sentinel Lymph Node Biopsy
Procedure: Axillary Dissection — Axillary dissection is the surgical removal of all Berg level I and II lymph nodes present in the axilla. The operation is carried out, at our Institute, during the surgery to treat the cancer in the breast (either breast-conserving surgery - quadrantectomy, or mastectomy).
  Other Names: Axillary Lymph Node Dissection
  Arms: SNB + AD

SUMMARY:
Many doctors believe that breast cancer patients scheduled for pre-operative chemotherapy whose cancer has spread to the axilla (determined by palpation plus ultrasound) should not receive sentinel node biopsy after chemotherapy, but proceed directly to removal of all the axillary lymph nodes.

In this study, breast cancer patients with operable medium-size cancer (T2) scheduled for pre-operative chemotherapy, and a disease-free or a metastatic axilla, are prospectively assigned to receive sentinel node biopsy as part of their post-chemotherapy surgical treatment (whose main aim is to remove the cancer in the breast).

Irrespective of whether the axilla is disease-free or metastatic before chemotherapy, if the removed sentinel nodes are disease-free on histological examination (pN0) after chemotherapy, then no further axillary treatment is given. If however the sentinel nodes contain cancer, then the other axillary lymph nodes will be removed surgically.

The study hypothesis is that, irrespective of whether the axilla is disease-free or metastatic before chemotherapy, patients with negative axillary sentinel nodes on histological examination (pN0) after chemotherapy, and who are no given further axillary treatment, will do as well as pN1 patients whose axillary lymph nodes are completely removed (a more aggressive treatment).

ELIGIBILITY:
Inclusion Criteria:

* cT2 cN0/1 breast cancer
* Scheduled for neoadjuvant chemotherapy,
* Informed consent,

Exclusion Criteria:

* Previous malignancy at another site
* Synchronous breast cancer at diagnosis
* Distant metastasis at diagnosis
* Clinically involved axilla (cN1) after neoadjuvant chemotherapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Yes
Enrollment: 353 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) and Disease-Free Survival (DFS) | Ten years
  DFS and OS are reckoned from date of surgery. DFS is time to recurrence or death, whichever occurred first. OS is time to death for any cause. Time is censored for living patients who are event-free at most recent follow up. OS and DFS curves are estimated using the Kaplan-Meier method and compared using the log-rank test. To compare DFS and OS in the SNB only and SNB + AD groups, propensity scores are estimated to account for bias due to non-random assignment to SNB vs SNB + AD

SECONDARY OUTCOMES:
Rate of axillary failure in those receiving only sentinel node biopsy | Ten years
  In patients given only sentinel node biopsy the proportion of patients who develop disease in the axilla will be calculated.

OTHER OUTCOMES:
Assessment of pathological response to primary chemotherapy as predictor of outcome | Ten years
  The response of the cancer to primary chemotherapy (complete response, partial response, stable disease, disease progression) will be related to overall outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Martelli, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano

IPD SHARING:
Plan to Share IPD: No